CLINICAL TRIAL: NCT02685800
Title: A Registry on Outcomes in Women Undergoing Assisted Reproductive Techniques After Recurrent Failures
Brief Title: Recurrent Failures in assIsted Reproductive Techniques (The FIRST Registry)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Casa Sollievo della Sofferenza IRCCS (Other)
Responsible Party: Principal Investigator, Elvira Grandone, MD, Head of Unit, Head of Unit, Casa Sollievo della Sofferenza IRCCS
Other Study IDs: FIRST - V 1_28 Ago 15
Record Dates: First submitted 2016-02-10; First posted 2016-02-19 (Estimated); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Months
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Assisted Reproductive Technologies (ARTs) are widely used in couples with fertility problems. However, despite ART treatment options have evolved over time, the implantation rate remains rather low.

A possible role for inherited and acquired thrombophilias has been invoked, especially in women with previous implantation failures. However, several factors could play a role in these conditions.

A potential benefit of low-molecular-weight heparin (LMWH) in improving ART outcomes, independently of the presence of thrombophilia, has been recently suggested.

This register is designed in order to better define all possible variables influencing ART outcome and improve clinical management of women with previous implantation failures. During this study the investigators will collect and evaluate clinical data regarding the first cycle in women with previous ART failures.

ELIGIBILITY:
Inclusion Criteria:

* 2 or more implantation failures/losses of clinical pregnancies after ART
* ART cycle at enrolment
* Informed consent

Exclusion Criteria:

* Ovarian hypofunction
* Uterine pathology
* Hydrosalpinges
* Previous inclusion in the study

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Consecutive women undergoing ART after recurrent failures.
Sampling Method: Probability Sample
Enrollment: 624 (Estimated)
Dates: Start 2015-10; Primary Completion 2020-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Number of live births | 10 months

SECONDARY OUTCOMES:
Number of clinical pregnancies after ART | 10 months

CONTACTS AND LOCATIONS:
Overall Officials: Elvira Grandone, Principal Investigator — IRCCS Casa Sollievo della Sofferenza - San Giovanni Rotondo, Foggia, Italy
Locations (1):
- IRCCS Casa Sollievo della Sofferenza, San Giovanni Rotondo, Foggia, Italy

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Villani M, Baldini D, Totaro P, Larciprete G, Kovac M, Carone D, Passamonti SM, Permunian ET, Bartolotti T, Lojacono A, Cacciola R, Pinto GL, Bucherini E, De Stefano V, Lodigiani C, Lavopa C, Cho YS, Pizzicaroli C, Colaizzo D, Grandone E. Rationale and design of two prospective, multicenter, observational studies on reproductive outcome in women with recurrent failures after spontaneous or assisted conception: OTTILIA and FIRST registries. BMC Pregnancy Childbirth. 2019 Aug 13;19(1):292. doi: 10.1186/s12884-019-2444-y. PMID 31409287